CLINICAL TRIAL: NCT01879943
Title: Capsule Versus Conventional Colonoscopy in Patient Following Colorectal Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Operational difficulties related to medical staff turnover (investigators departure and sickness leave).
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 12-003; 2012-A01475-38 (Other: ANSM France)
Record Dates: First submitted 2013-06-14; First posted 2013-06-18 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Follow up; Colonoscopy; Videocapsule
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- PillCam COLON 2 and Standard Colonoscopy (Experimental): Patients will have videocapsule colonoscopy after bowel preparation, followed by standard colonoscopy the next day.
  Interventions:
  * Device: PillCam COLON 2 on D0
  * Procedure: Standard colonoscopy on D1
  Interventions: Device: PillCam Colon 2; Procedure: Colonoscopy

INTERVENTIONS:
Device: PillCam Colon 2 — PillCam® COLON 2 capsule endoscopy is a minimally invasive tool for direct visualization of the colon, including identifying the occurrence of polyps.
Procedure: Colonoscopy — Standard colonoscopy is the standard against which capsule endoscopy is compared.

SUMMARY:
The study will compare the diagnostic efficacy of the VCC (PillCam COLON 2) to standard colonoscopy in patients with prior colorectal surgery.

The hypothesis is to validate the VCC as a means of screening for colonic polyps after resection, which would avoid a colonoscopy with its associated general anesthesia and potential side effects.

DETAILED DESCRIPTION:
Standard care after colorectal surgery is colon surveillance by standard colonoscopy with its benefits (gold standard examination, resection of lesions) and disadvantages (acceptability, general anesthesia, availability of qualified personnel, risk of perforation and associated gastrointestinal bleeding).

Use of a video-capsule (VCC) is a new, non-invasive technique, that allows to visualize the colon as a whole. This technique has the advantage of not requiring general anesthesia or air insufflation. The examination is performed as an outpatient procedure and therefore does not require hospitalization.

In previous studies, PillCam COLON 2 showed a good sensitivity and specificity in detecting colorectal lesions. However, its use requires an excellent bowel preparation.

To date, no study has been conducted using the VCC in monitoring patients with prior colorectal surgery, especially on the passage of the VCC through surgical anastomosis. No information on VCC capabilities to view and recognize surgical anastomoses and VCC transit time in surgically modified colon is available. The possibility to precisely locate a colorectal lesion prior to surgery, using the VCC, also remains to be studied.

The study requires a 2-month patient participation. The planned total study duration is 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. patient between 18 and 85 years old
2. patient with greater than 3 month follow-up for colorectal resection with ileo-colic , colo-colic or colorectal anastomosis, regardless of etiology
3. patient requiring a colonoscopy for regular medical care
4. absence of contra-indication to anesthesia and to colonoscopy conduct
5. patient able to understand the study related information and to provide written informed consent
6. patient registered with the French social security regime

Non-inclusion Criteria:

1. absence of written informed consent
2. patient having had a total colectomy
3. patient with terminal stoma
4. patient with clinical suspicion of intestinal stenosis and/or anastomotic stenosis
5. patient with known Zenker diverticulum
6. patient wearing a pacemaker or any other internal electronic medical device
7. patient with deglutition disorders and/or altered state of consciousness
8. patient with serious disease preventing planned study procedures
9. pregnant or breast-feeding woman
10. patient within exclusion period from other clinical trial
11. patient having forfeited their freedom of an administrative or legal obligation
12. patient being under guardianship

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-10-18 (Actual); Primary Completion 2016-06-08 (Actual); Study Completion 2016-06-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with full colonic exploration and detection of lesions | By the end of both procedures (Day 1)
  Number of patients for whom the capsule allowed for full colonic exploration and presence/absence of colorectal lesions detected by VCC compared to conventional colonoscopy

SECONDARY OUTCOMES:
Anastomosis visualization | Prior to colonoscopy on Day 1
  Anastomosis visualization by VCC and type (latero-lateral, termino-lateral, latero-terminal and termino-terminal)
Number and size of detected lesions | By the end of both procedures (Day 1)
  Number and size of detected lesions with VCC compared to conventional colonoscopy
Quality of colic preparation | By the end of both procedures (Day 1)
  Assessment of the quality of colic preparation for VCC (D0) and colonoscopy (D1)
Times related to videocapsule | Prior to colonoscopy on Day 1
  Assessment of times related to videocapsule:
  * Transit time of videocapsule : from ingestion to expulsion
  * Reading time : time required for reading and analysing videocapsule recordings by gastroenterologist
Adverse events related to VCC exam and colonoscopy | Until end of Day 1
  Assessment of safety of each method. Recording of adverse events.
Patient's assessment of tolerability and acceptance | Follow up visit (between Day 15 and Day 30)
  Patient ranking of tolerability and acceptance of each of the procedures using a visual analog scale
Health-economic assessment | End of follow-up (between D15 and D30)
  Assessment of costs associated to each of the exams:
  * Colonoscopy duration (OR entry - exit)
  * Device cost (coloscope, capsule)
  * Cost of medical exams related to each procedure (from pre-anesthesia to follow-up)
  * Cost of medical time related to each procedure

CONTACTS AND LOCATIONS:
Overall Officials: Michel Delvaux, MD, Principal Investigator — Department of Hepato-Gastroenterology, Nouvel Hopital Civil, Strasbourg, France
Locations (1):
- Department of Hepato-Gastroenterology, Nouvel Hopital Civil, Strasbourg, France